CLINICAL TRIAL: NCT06612021
Title: Clinical Performance of Posterior Restorations Using Hema Free Universal Adhesive Versus Hema Containing Universal Adhesive Over One Year Using USPHS Criteria: Randomized Controlled Trial
Brief Title: Hema Free Versus Hema Containing Adhesives in Posterior Restorations
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Fathi Abdelsalam, lecturer of conservative dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2255874
Record Dates: First submitted 2023-08-25; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Dental Caries
Keywords: HEMA free; HEMA containing adhesive; Giomers; Giomer; USPHS criteria
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HEMA free universal adhesive group (Experimental)
  Interventions: Procedure: Beautibond universal adhesive
- HEMA containing universal adhesive group (Active Comparator)
  Interventions: Procedure: Tetric N universal bond

INTERVENTIONS:
Procedure: Beautibond universal adhesive — HEMA free universal adhesive
  Arms: HEMA free universal adhesive group
Procedure: Tetric N universal bond — HEMA containing universal bond
  Arms: HEMA containing universal adhesive group

SUMMARY:
The aim of study is to evaluate the clinical performance of posterior restorations using HEMA free universal adhesive versus HEMA containing universal adhesive over one year using USPHS criteria.

DETAILED DESCRIPTION:
The study is intended to evaluate the HEMA free universal adhesive versus HEMA containing universal adhesive when both used in conjunction with giomer aesthetic restorations in occlusal cavities in posterior teeth ICDAS III and IV.

The restorations will be evaluated at baseline, 6 and 12 months according to modified USPHS criteria in terms of marginal staining, marginal adaptation and caries recurrence.

Patients will be recruited from outpatient clinic of conservative dentistry department, cairo university according to inclusion and exclusion criteria. patient will be randomly allocated to intervention or control group.

ELIGIBILITY:
Inclusion Criteria of participants:

* Patients with occlusal caries in molars classified as ICDAS III or IV.
* 19-35 years.
* Males or Females.
* Co-operative patients approving to participate in the trial.

Exclusion criteria of participants:

* Pregnancy.
* Disabilities.
* Systemic disease or severe medical complications.
* Allergic history concerning methacrylate.
* Rampant caries.
* Heavy smoking.
* Xerostomia.
* Lack of compliance.
* Evidence of severe bruxism, clenching, or tempromandibular joint disorders.

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2024-10-14 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
marginal staining of restoration | baseline ,6 months & 12 months
  marginal staining using USPHS criteria Alpha: No staining in the margin Bravo: superficial staining on the margin Charlie: deep staining on the margin

SECONDARY OUTCOMES:
caries recurrence | baseline ,6 months ,12 months
  caries recurrence using USPHS criteria Alpha: no recurrent caries Charlie: Caries recurrence
marginal adaptation of restoration | baseline ,6 months and 12 months
  marginal adaptation using USPHS criteria ALPHA: Marginal continuity BRAVO: slightly detectable marginal discontinuity that does not require replacement CHARLIE: Detectable crevice or ledge at margin that requires replacement

CONTACTS AND LOCATIONS:
Overall Officials: Alaa F Abdelsalam, phD, Principal Investigator — lecturer of conservative dentistry, Cairo university; Hadier M Gad, PhD, Principal Investigator — Lecturer of conservative dentistry, Cairo university; Manar A Elmokanen, PhD, Principal Investigator — Lecturer of conservative dentistry, Cairo University
Locations (1):
- Faculty of dentistry Cairo university, Cairo, Manyal, Egypt

IPD SHARING:
Plan to Share IPD: No